CLINICAL TRIAL: NCT07134309
Title: Comparison of the Effectiveness of Mat Pilates and Reformer Pilates on Pain, Functional Disability and Quality Of Life in Women With Non-Specific Low Back Pain: A Randomized Controlled Study
Brief Title: Comparison of the Effectiveness of Mat Pilates and Reformer Pilates in Women With Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-471
Record Dates: First submitted 2025-08-12; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Low Back Pain
Keywords: reformer pilates; mat pilates; posture exercises; pain; functional disability; quality of life
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomised controlled trial. One group received reformer Pilates training, another group received mat Pilates training, and the third group received posture exercises.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Instrumental Pilates (Experimental): Instrumental pilates group received reformer Pilates for 12 weeks.
  Interventions: Other: Exercise Training
- Mat Pilates (Experimental): Mat pilates group received mat Pilates training for 12 weeks.
  Interventions: Other: Exercise Training
- Posture Exercises (Experimental): The third group received posture exercise training for 12 weeks
  Interventions: Other: Exercise Training

INTERVENTIONS:
Other: Exercise Training — Reformer, mat pilates, and general posture exercise training were performed twice a weekly for 12 weeks. Before starting pilates training, the key elements of pilates were taught to patients for one session. In evaluation, Visual Analog Scale (VAS) was used for pain intensity, Oswestry Low Back Pain Questionnaire for disability, Short Form - 36 Questionnaire (SF-36) for quality of life, Sit-lie test for flexibility, McGill extension test for trunk extension endurance. Demographic information of individuals was recorded.
  Other Names: Pilates and posture exercises

SUMMARY:
In this study, the effects of instrumental pilates, mat pilates and general posture exercises on pain, disability, quality of life, flexibility and endurance of trunk extension muscles were researched in women with non-specific low back pain. The aim of this study was to examine the superiority of exercises over each other.

DETAILED DESCRIPTION:
The participants were divided into three groups as reformer pilates group, mat pilates group and control group. Patients were allocated to the groups according to order of arrival starting from the reformer pilates group using a simple basic randomization method. All assessments were performed face to face by the physiotherapist. Exercise follow-up was performed individually. Pain intensity, level of disability, flexibility values, quality of life, and trunk extension endurance times were evaluated before and after treatment. Reformer, mat pilates, and general posture exercise training were performed twice a weekly for 12 weeks. In evaluation, Visual Analog Scale (VAS) was used for pain intensity, Oswestry Low Back Pain Questionnaire for disability, Short Form - 36 Questionnaire (SF-36) for quality of life, Sit-lie test for flexibility, McGill extension test for trunk extension endurance. Demographic information of individuals was recorded.

ELIGIBILITY:
Inclusion Criteria:

* being a woman between the ages of 18 and 50
* having a diagnosis of NLBP
* not having any obstacles to exercise.

Exclusion Criteria:

* To be pregnant, history of previous spine surgery, rheumatic diseases that may cause low back pain, severe spinal pathologies (tumor, fracture, etc.).
* having received physiotherapy for spine health in the last 6 months and receiving any analgesic or anti-inflammatory medical treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Disability | baseline and after 12 weeks training immediately after the intervention
  Oswestry Low Back Pain Questionnaire: There are 10 subheadings in this Questionnaire.There are six options under each heading.In each section, options are scored between 0-5.The lowest score obtained as a result of the survey is "0" and the highest score is "50". The level of functional disability increases with increasing total score.
Pain Level | baseline and after 12 weeks training immediately after the intervention
  Visual Pain Scale: '0' indicates no pain, '10' indicates severe pain. As the score increases, the level of pain worsens.
Flexibility | baseline and after 12 weeks training immediately after the intervention
  Sit and Reach test: A test box with a ruler was used. The participants placed their feet on the corners of the box without shoes.The data was recorded in centimetres. The corner of the test box is considered to be 0,Values extending further from the edge of the cube were accepted as positive, while values beyond were accepted as negative .
Quality of Life Level | baseline and after 12 weeks training immediately after the intervention
  Short Form-36 Questionnaire: It has 8 subscales of health- related quality of life that examine physical functioning (10 items). Each subscale is calculated separately. In the questionnaire, a minimum of 0 and a maximum of 100 points are awarded.. A score of '0' indicates poor health, while a score of '100' indicates good health.
Trunk Extension Endurance | baseline and after 12 weeks training immediately after the intervention
  The McGill trunk extension test: The time the individuals were able to maintain the position was recorded in seconds.Minimum and maximum values depend on participants.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Kübra AY, RA, Principal Investigator — Ankara Yildirim Beyazıt University; Bahar ANAFOROĞLU, PROF, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No